CLINICAL TRIAL: NCT06729502
Title: Pictorial Fit-Frail Scale in Adults Admitted to the Intensive Care Unit in a Tertiary Center- an Observational Prospective Study
Brief Title: Pictorial Fit-Frail Scale in Adults Admitted to the ICU in a Tertiary Center- an Observational Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Liran Statlender, Senior Physician, principal investigator, Rabin Medical Center
Other Study IDs: 0377-24-RMC
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-12

CONDITIONS: Frail

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire - Pictorial Fit-Frail Scale — All patients over 60 years old, or their caregivers, will be asked to fill the PFFS questionnaire

SUMMARY:
Understanding the frailty levels of critically ill patients using the PFFS at time of admission to ICU.

Exploring any associations between frailty, other prognostic factors, and patient outcomes.

DETAILED DESCRIPTION:
Frailty is a state of high vulnerability for adverse health outcomes, including disability, dependency, falls, need for long-term care, and mortality. Several definitions exist, but all measure one's vulnerabilities, strengths, and indirectly assess the physiological reserve. Frailty is not necessarily age dependent, but some of its domain are affected by age. In recent years, frailty has increasingly been recognized as an important factor in the prognosis assessment of an older critically ill patient, in terms of mortality (both in-hospital and long term), hospital length of stay (LOS) and discharge disposition. A previous study performed in Rabin Medical Center ICU demonstrated a strong association between frailty in 90-d mortality of critically ill patients. Frailty is also associated with a higher risk of persistent clinical illness (critical care dependency for survival).

There are several methods for frailty assessment; the comprehensive geriatric assessment is considered the gold standard. However, this method takes time, and requires full patient cooperation, both are usually not possible at the time of critical illness. Several other valeted methods are commonly used, including the Clinical Frailty Scale (CFS), Frailty Index, Frailty phenotype, simple FRAIL questionnaire modified frailty index, and many more.These tools have been validated in different settings, and were found related to several outcomes. There are several differences between the different tools. Some require clinical assessment (with or without patients cooperation), while others require only a review of the healthcare record (EHR). Nevertheless, there are differences between these tools in sensitivity, and specificity in terms of screening and diagnosis of frailty and the contributing factors to the state of frailty.

In 2019 the pictorial fit-frail scale (PFFS) has been introduced as a quick and easy-to-use tool for frailty assessment. It takes few minutes to fill by the patient or caregiver, it's not based on language or health literacy, and requires no clinical examination by the medical staff. The PFFS was validated in several clinical settings, including thoracic surgery clinic, geriatric clinic, memory clinic, and primary care clinics.

PFFS has been assessed in the critical care setting in our unit and was found associated with longer term mortality. The PFFS questionnaire has become a standard of care upon admission to our ICU. This study aims to describe the PFFS scores patients over 60 years old, its correlation with other prognostic scores, and its association with patients' outcomes (ICU length of stay, length of ventilation, ICU mortality, 90days mortality).

ELIGIBILITY:
Inclusion Criteria:

* Older adults (age ≥ 60 years) who were admitted to the ICU for more than 24 hours at the participating centers

Exclusion Criteria:

* Prior recent admission to an ICU (within 30 days)
* Admissions for brain death evaluation.
* Planned admissions to the ICU (i.e for percutaneous tracheostomy, for specific treatment under sedation).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 60 years old or more who admitted to the ICU for more than 24 hours, for any reason (except from those specified in the exclusion criteria)
Sampling Method: Non-Probability Sample
Enrollment: 1350 (Estimated)
Dates: Start 2025-01-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
90-d mortality | up to 90 days from ICU admission
  Mortality at 90 days from ICU admission

SECONDARY OUTCOMES:
ICU mortality | During index admission
  Mortality during index admission at the ICU
Hospital mortality | During index admission
  Mortality during hospital admission
ICU length of stay | up to 90 days from ICU admission
  Duration of ICU admission
Hospital length of stay | Up to 90 days from ICU admission
  Duration of hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No